CLINICAL TRIAL: NCT01092481
Title: A Randomized Phase III Study Investigating the Role of Oxaliplatin Duration (3 Months Versus 6 Months) in Modified FOLFOX-6 or CAPOX Regimen as Adjuvant Therapy for Patients With Stage II/III Colon Cancer
Brief Title: Study Investigating the Role of Oxaliplatin Duration in Modified FOLFOX-6 or CAPOX Regimen as Adjuvant Colon Cancer Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Suk Park, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-11-008; 2009-11-008 (Other: Samsung Medical Center)
Record Dates: First submitted 2009-11-22; First posted 2010-03-25 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Colon Cancer
Keywords: Adjuvant FOLFOX or CAPOX Therapy; Stage II/III Colon Cancer; Adjuvant Therapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFOX_12 or CAPOX_8 (Active Comparator): 6 months of oxaliplatin in 12 cycles of modified FOLFOX-6 or 8 cycles of CAPOX
  Interventions: Drug: oxaliplatin
- FOLFOX_6 or CAPOX_4 (Experimental): 3 months of oxaliplatin in 12 cycles of modified FOLFOX-6 or 8 cycles of CAPOX
  Interventions: Drug: oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin — to confirm that first 3 months of oxaliplatin in 12 cycles of modified FOLFOX-6 or 8 cycles of CAPOX treatment is not inferior to 6 months of oxaliplatin in modified FOLFOX-6 or CAPOX treatment in terms of disease free survival in patients with stage II/III colon cancer.
  Other Names: oxaliplatin (modified FOLFOX-6 OR CAPOX)

SUMMARY:
This study is designed to confirm that first 3 months of oxaliplatin in 6 months of modified FOLFOX-6 or CAPOX treatment is not inferior to 6 months of oxaliplatin in modified FOLFOX-6 or CAPOX treatment in terms of disease free survival in patients with stage II/III colon cancer.

DETAILED DESCRIPTION:
This study is designed to confirm that first 3 months of oxaliplatin in 6 months of modified FOLFOX-6 or CAPOX treatment is not inferior to 6 months of oxaliplatin in modified FOLFOX-6 or CAPOX treatment in terms of disease free survival in patients with stage II/III colon cancer. In addition, we would like to characterize pharmacogenomic profile associated with toxicities and gene expression profiling to predict the recurrence of colon cancer as parallel study.

ELIGIBILITY:
Inclusion Criteria:

* Curatively resected, histologically confirmed colon adenocarcinoma
* AJCC/UICC high-risk stage II, stage III colon cancer
* Age over 18 years old
* Performance status (ECOG scale): 0-1
* Adequate major organ functions
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Colon cancer other than adenocarcinoma
* Rectal cancer
* R1 or R2 resections
* Other malignancies within the last 5 years
* Symptomatic peripheral sensory neuropathy
* Presence of other serious disease
* Lactating or pregnant women
* Fertile women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1580 (Actual)
Dates: Start 2010-01-26 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years
quality of life | 3 years
safety profiles | 3 years
  Safety will be assessed on the basis of an analysis of adverse events, standard clinical chemistry and hematology findings. Clinical and laboratory toxicities/symptoms will be graded according to the CTCAE 3.0. Adverse events which are not reported in CTCAE 3.0 will be graded as mild, moderate, severe or life threatening.

CONTACTS AND LOCATIONS:
Overall Officials: Young Suk Park, M.D.,Ph.D., Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (17):
- South Korea (17):
  - Hallym University Medical Center, Anyang-si, Gyeonggi-do
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - School of Medicine, CHA University, Seongnam-si, Gyeonggi-do
  - Sungkyunkwan University Masan Samsung Hospital, Masan, Gyeongsangnam
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam
  - Kosin Medical Center, Busan
  - Dong-A University Medical Center, Busan
  - Gachon University Gil Hospital, Incheon
  - Yonsei University College of Medicine, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's hospital, Catholic Univerisity, Seoul
  - Asan Medical Center, Seoul
  - Soonchunhyang University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Chung-Ang University College of Medicine, Seoul

REFERENCES:
- [Derived] Kim ST, Kim SY, Lee J, Yun SH, Kim HC, Lee WY, Kim TW, Hong YS, Lim SB, Baek JY, Oh JH, Ahn JB, Shin SJ, Han SW, Kim SG, Kang SY, Sym SJ, Zang DY, Kim YH, Choi IS, Kang JH, Kim MJ, Park YS. Oxaliplatin (3 months v 6 months) With 6 Months of Fluoropyrimidine as Adjuvant Therapy in Patients With Stage II/III Colon Cancer: KCSG CO09-07. J Clin Oncol. 2022 Nov 20;40(33):3868-3877. doi: 10.1200/JCO.21.02962. Epub 2022 Jun 30. PMID 35772045